CLINICAL TRIAL: NCT05045170
Title: The Influence of Propofol and Dexmedetomidine Sedation on Memory Consolidation
Brief Title: Sedation and Memory Consolidation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: I.M. Sechenov First Moscow State Medical University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Basic Science
Other Study IDs: 2107
Record Dates: First submitted 2021-09-06; First posted 2021-09-16 (Actual); Last update posted 2022-02-09 (Actual); Status verified 2021-07

CONDITIONS: Memory Impairment; Amnesia; Recall; Recognition
Keywords: sedation; Memory consolidation; Propofol; Dexmedetomidine
MeSH Terms: conditions — Memory Disorders; Amnesia

STUDY DESIGN:
Who Masked: Participant
Masking Description: Participants were not aware of the drug used for sedation
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- propofol group (Experimental): patients with American Society of Anesthesiologists (ASA) I-II, Montreal cognitive assessment test≥26, trauma surgery under spinal anesthesia with propofol sedation
  Interventions: Drug: Influence of propofol sedation on memory consolidation and 'working memory'
- dexmedetomidine group (Experimental): patients with American Society of Anesthesiologists (ASA) I-II, Montreal cognitive assessment test≥26, trauma surgery under spinal anesthesia with dexmedetomidine sedation
  Interventions: Drug: Influence of dexmedetomidine sedation on memory consolidation and 'working memory'
- control group (Placebo Comparator): patients with American Society of Anesthesiologists (ASA) I-II, Montreal cognitive assessment test≥26, trauma surgery under spinal anesthesia without sedation
  Interventions: Drug: Influence of spinal anesthesia on memory consolidation and 'working memory'

INTERVENTIONS:
Drug: Influence of propofol sedation on memory consolidation and 'working memory' — Spinal anesthesia is performed by anesthesiologist. Memory testing is conducted immediately prior to propofol sedation (stage 1), 5-10 minutes after the start of propofol sedation (stage 2), 10 minutes after propofol sedation is finished and consciousness is restored (stage 3). Five emotionally neutral words are heard by the patients twice at each stage to assess the impact of sedation on memory consolidation. The patients repeat the memorized words after each audition. To assess the effect of sedation on the 'working memory', anesthesiologist asked the patient to remember and reproduce the memorized words five minutes after learning in the second stage. Approximately, 24 hours after the end of anesthesia, recall and recognition of the experimental words are tested. The number of words in recall and recognition testing is recorded by researcher.
  Arms: propofol group
Drug: Influence of dexmedetomidine sedation on memory consolidation and 'working memory' — Spinal anesthesia is performed by anesthesiologist. Memory testing is conducted immediately prior to dexmedetomidine sedation (stage 1), 5-10 minutes after the start of dexmedetomidine sedation (stage 2), 10 minutes after dexmedetomidine sedation is finished and consciousness is restored (stage 3). Five emotionally neutral words are heard by the patients twice at each stage to assess the impact of sedation on memory consolidation. The patients repeat the memorized words after each audition. To assess the effect of sedation on the 'working memory', anesthesiologist asked the patient to remember and reproduce the memorized words five minutes after learning in the second stage. Approximately, 24 hours after the end of anesthesia, recall and recognition of the experimental words are tested. The number of words in recall and recognition testing is recorded by researcher.
  Arms: dexmedetomidine group
Drug: Influence of spinal anesthesia on memory consolidation and 'working memory' — Spinal anesthesia is performed by anesthesiologist. Memory testing is conducted immediately prior to operation (stage 1), 5-10 minutes after the start of operation (stage 2), 10 minutes before the end of operation (stage 3). Five emotionally neutral words are heard by the patients twice at each stage to assess the impact of sedation on memory consolidation. The patients repeat the memorized words after each audition. To assess the effect of sedation on the 'working memory', anesthesiologist asked the patient to remember and reproduce the memorized words five minutes after learning in the second stage. Approximately, 24 hours after the end of anesthesia, recall and recognition of the experimental words are tested. The number of words in recall and recognition testing is recorded by researcher.
  Arms: control group

SUMMARY:
The study of plasticity processes, in particular, memory, is one of the fundamental directions in anesthesiology. To date, there are different views on the impact of sedation and anesthesia on memory. Memory consolidation is one of the most crucial processes that the anesthesiologist is interested in. Memory consolidation is the mechanism of transferring short-term memory to long-term memory. The investigators suppose that propofol or dexmedetomidine sedation disrupts memory consolidation. In addition, the investigators inquired about the impact of sedation on 'working memory'. Therefore, a better understanding of the influence of anesthesia and sedation on basic memory processes will allow the anesthesiologist to balance the choice of the drug and ensure the patient's safety in the intraoperative period.

DETAILED DESCRIPTION:
The study is a prospective, randomized, single blind design. Patients undergoing elective trauma surgery (arthroscopy, reconstructive foot surgery) under subarachnoidal anesthesia are enrolled in this study. All patients were randomly divided into three groups depending on the drug type: first - propofol, second - dexmedetomidine, third - control.

The Montreal cognitive assessment test (MoCA - test) is a high validity test. MoCA - test is used to determine cognitive impairments in patients in the pre-operative period. The MoCA test time is approximately 10 minutes. The maximum possible score is 30; 26 points and more are considered normal, 25 or less is evidence of cognitive impairment.

American Society of Anesthesiologists (ASA) physical status classification system is used to assess and communicate a patient's pre-anesthesia medical co-morbidities (ASA I - a normal healthy patient, ASA II - a patient with mild systemic disease, ASA III - a patient with severe systemic disease, ASA IV - a patient with severe systemic disease that is a constant threat to life, ASA V - a moribund patient who is not expected to survive without the operation, ASA VI - a declared brain-dead patient whose organs are being removed for donor purposes.

To determine the level of anxiety and depression in the preoperative period, patients are tested using the Hospital Anxiety and Depression Scale (HADS). Values on the HADS scale<7 points are interpreted as normal, with scores from 8 to 10 as subclinically expressed anxiety and/or depression, and above 10 points-clinically expressed anxiety and/or depression.

In the operating room intravenous (i.v.) peripheral canulla Vasofix Certo (B. Braun, Germany) with a diameter of 18 or 20 Gauge is inserted before the start of regional anesthesia for infusion therapy. Before spinal anesthesia an anesthesiologist inject 0.9% saline infusion (Grotex, Russia) of 6-8 ml/kg.

Following this procedure, the investigators perform a puncture of the subarachnoid space with a 27 Gauge Pencil Point needle (Bbraun, Germany) under aseptic conditions under local anesthesia with lidocaine (Pharmasyntez, Russia) at the L2-L4 level. The criterion for verifying the subarachnoid space is the appearance of liquor in the needle pavilion. After performing the aspiration test, 10-15 mg of an isobaric solution of moxicaine (Novosibhimfarm, Russia) is injected. To evaluate the sensory block, the investigators use the tactile sensitivity loss test ('pinprick' test), and the motor block-the Bromage test.

0.9% saline (20 - 25 ml/kg) is administered to patients in the all groups. Propofol (1 group (Propofol Kabi, Registration number from the State Register of Medicines - 000875)) or dexmedetomidine (2 group (Dexmedetomidine, Registration number from the State Register of Medicines - 005916) are used for sedation. Intravenous infusion of propofol or dexmedetomidine is performed with a BBraun Space (B. Braun Melsungen AG, Registration certificate for a medical device RZN 2013/905). Target control infusion (TCI, Shnider model) is applied for the dosing of propofol concentration. At the beginning of sedation, the level of the target propofol concentration is 1.5 - 2 mcg ml-1, during operation - 2.5 mcg ml-1. Intravenous infusion of dexmedetomidine starts with a dose of 1 mcg/kg for 10 minutes, with maintaining dose from 0.6 to 0.7 mcg/kg/min follows by titration from 0.2 to 2 mcg/kg/h depending on the level of sedation. Propofol or dexmedetomidine infusion terminates 10 minutes before the end of the operation. 0.9% saline (20 - 25 ml/kg) is administered to patients in the control group (3 group). Sedation is not performed in control group.

The Richmond agitation and sedation Scale (RASS) and bispectral index monitor A-2000XP (BIS, Aspect Medical Systems, Inc. (USA), Registration certificate for a medical device RZN 2005/498) are used to assess the depth of sedation. RASS values '-2' - '-3' (short-term eyes opening for less than 10 seconds or voluntary movements without eye contact in response to a call) correspond to light-moderate sedation, '-4' (eyes opening or voluntary movements in response to physical stimulation) - deep sedation. BIS values 70 - 90 correspond to light - moderate sedation, 60 - 70 - deep sedation.

To ensure patient safety, the investigators use the basic monitoring standard: noninvasive arterial pressure (NAP), heart rate (HR), electrocardiogram (ECG), SpO2, capnography (Philips Monitor IntelliVue MP40 (Medizin Systeme Boblingen GmbH, Germany, Registration certificate for a medical device RZN 2014/2009)).

Memory testing is conducted in three stages. Stage 1 - immediately prior to sedation, stage 2 - 5-10 minutes after the start of sedation (RASS '-1' - '-2', BIS 70 - 90), stage 3 - 10 minutes after sedation is finished and consciousness is restored (RASS '0', BIS 95 - 100). Five emotionally neutral words are heard by the patients twice at each stage to assess the impact of sedation on memory consolidation. The experimental words are different at each stage. The patients repeat the memorized words after each audition. To assess the effect of sedation on the 'working memory', anesthesiologist asked the patient to remember and reproduce the memorized words five minutes after learning in the second stage. Approximately, 24 hours after the end of anesthesia, recall and recognition of the experimental words are tested. To assess recall, the patients remember all the words listened before, during and after anesthesia. To test recognition, patients use to mark the words learned during surgery in the list of words, which consists of 15 experimental and 10 control. The number of words in recall and recognition testing is recorded by researcher.

Statistical analysis is perfomed in MS Excel and Jamovi 2.0.0 programs. The Shapiro-Wilk and Kolmogorov-Smirnov tests are used to determine the normality of the distribution. The analysis of the categorical variables is evaluated using the criterion χ2. For inter-group comparison of quantitative variables, one-way analysis of variance (one-way ANOVA) followed by post-hoc Bonferroni test are used. Repeated measures analysis of variance (RM-ANOVA) followed by post hoc tests for multiple comparisons, which are Bonferroni-adjusted, are performed to compare data within groups. Statistical significance level is set at P < 0.05.

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent
* Age ≥ 18 and ≤70 years
* Elective trauma surgery (arthroscopy, reconstructive foot surgery) under regional anesthesia (spinal anesthesia) with propofol, dexmedetomidine or without sedation
* Montreal cognitive assessment test ≥ 26
* Patients with American Society of Anesthesiologists (ASA) I-II

Non-inclusion criteria:

* Not written informed consent to participate in the research and/or perform regional blockade
* Age˂18 and ˃70 years
* Allergy to propofol, dexmedetomidine, lidocaine, bupivacaine
* Pregnancy
* Epilepsy anamnesis
* II-III degree atrioventricular block
* Montreal cognitive assessment test ˂ 26
* Patients with American Society of Anesthesiologists (ASA) ˃ II
* Emergency operation
* The presence of psychiatric disorders
* Сancer patients with a life expectancy of less than two years
* Taking anticoagulants, psychotropic drugs

Exclusion Criteria:

* Patient refuse from further participation
* Ineffective spinal anesthesia
* Allergy on anesthesia drugs during perioperative period

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 81 (Actual)
Dates: Start 2021-05-11 (Actual); Primary Completion 2022-01-13 (Actual); Study Completion 2022-01-13 (Actual)

PRIMARY OUTCOMES:
memory consolidation impairment with propofol sedation | 24 hours after the end of anesthesia
  Memorizing emotionally neutral words before, during and after propofol sedation. Evaluation of recall and recognition of words 24 hours after anesthesia.
memory consolidation impairment with dexmedetomidine sedation | 24 hours after the end of anesthesia
  : Memorizing emotionally neutral words before, during and after dexmedetomidine sedation. Evaluation of recall and recognition of words 24 hours after anesthesia.
memory consolidation impairment without sedation | 24 hours after the end of anesthesia
  Memorizing emotionally neutral words before, during and after operation. Evaluation of recall and recognition of words 24 hours after anesthesia.

SECONDARY OUTCOMES:
'working memory' impairment with propofol sedation | 5 minutes after memorizing emotionally neutral words during propofol sedation
  Memorizing emotionally neutral words during propofol sedation (stage 2). Evaluation of remembering and reproducing of words five minutes after learning.
'working memory' impairment with dexmedetomidine sedation | 5 minutes after memorizing emotionally neutral words during dexmedetomidine sedation
  Memorizing emotionally neutral words during dexmedetomidine sedation (stage 2). Evaluation of remembering and reproducing of words five minutes after learning.
'working memory' impairment without sedation | 5 minutes after memorizing emotionally neutral words during operation
  Memorizing emotionally neutral words during operation (stage 2). Evaluation of remembering and reproducing of words five minutes after learning.

CONTACTS AND LOCATIONS:
Overall Officials: Vyacheslav Churakov, PgS, Principal Investigator — I.M. Sechenov First Moscow State Medical University (Sechenov University)
Locations (1):
- City Clinical Hospital № 31 of the Department of Health of Moscow, Moscow, Russia

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol, SAP, ICF
Time Frame: The data will become available 31.10.2021

REFERENCES:
- See also: Related Info — https://lomonosov-msu.ru/archive/Lomonosov_2020/data/19419/112756_uid128092_report.pdf
- See also: Related Info — https://istina.msu.ru/conferences/presentations/327241590/
- See also: Related Info — https://istina.msu.ru/publications/article/352671421/